CLINICAL TRIAL: NCT04856462
Title: The Alzheimer's Companion Engagement (ACE) Project.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sheria Robinson-Lane, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00230940; 1K01AG065420-01A1 (NIH)
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Stress, Psychological; Adaptation, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to intervention groups where they will receive structured education and support.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregiver Support (Experimental): All participants in all groups will receive 6 weeks of caregiving support including a weekly video/teleconference call, and handouts covering relevant educational topics)
  Interventions: Behavioral: Education Support

INTERVENTIONS:
Behavioral: Education Support — Caregivers engage in a weekly video/teleconference support group with a skilled facilitator to discuss various strategies for managing caregiving stress, challenging behaviors, and personal self-care.

SUMMARY:
Black family caregivers of older adults with Alzheimer's disease and/or related dementias (ADRD), have an increased mortality risk related to pre-existing health conditions and stress. Targeted, culturally responsive, health interventions that help Black ADRD caregivers to effectively manage their own health and use community preferenced ways of coping, can improve caregivers' overall health, perceived ability to provide care for a person with ADRD (self-efficacy), and increases the likelihood that they will experience benefits from caregiving. This clinical trial pilot will test the feasibility of a community based intervention designed to improve health outcomes for Black family caregivers of persons with ADRD.

DETAILED DESCRIPTION:
The proposed intervention is a peer-supportive and facilitator-led video teleconference program that will engage small groups of caregivers weekly over 6 weeks. Each week participants (n = 36, 2-5/group) will receive a different culturally relevant caregiving or personal health strategy to practice. During the support calls, a facilitator will provide an overview of the content covered and each participant will have the opportunity to discuss their past week and how they engaged the weekly strategy, or challenges that came up for them during the week. The format will be structured to ensure that core content is reviewed, and everyone can be equally engaged while flexible enough that caregivers can receive support in the areas they need. A battery of assessment measures will be taken at weeks 1 and 8.

ELIGIBILITY:
Inclusion criteria for participation are as follows:

Self-identified as Black/ African American At least 18 years old Able to speak, understand, and hear spoken English Related to, or has a close personal relationship to a person over the age of 55 that has an ADRD diagnosis or evidence of cognitive impairment Regular access to a smartphone, tablet or computer with internet access that will allow video conferencing engagement.

Provides monitoring, and assistance in activities of daily living and or other care tasks for the care recipient.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Caregiver Self-efficacy | 6 weeks
  Caregiver self-efficacy will be measured by the Revised Scale for Caregiving Self-Efficacy, which evaluates the caregivers' ability to obtain respite care, respond to disruptive behaviors, and control one's own upsetting thoughts about caregiving.

SECONDARY OUTCOMES:
Positive Aspects of Caregiving | 6 weeks
  Positive Aspects of Caregiving will be an additional outcome measure. The Positive Aspects of Caregiving tool is a brief tool that asks questions about caregiving experiences that made the caregiver feel good about providing care.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that the following data will be generated and made available 1) published tables, figures, graphs, and tables of data used for making graphs; 2) published journal papers, conference papers, annual reports and the final report; and 3) educational materials resulting from intervention development. All data will conform with relevant data and terminology standards.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: No less than 5 years following the date of the project completion or the date of study publication.
Access Criteria: To facilitate data sharing, project data will be made publicly available via a university-managed repository Deep Blue.
URL: http://deepblue.lib.umich.edu